CLINICAL TRIAL: NCT03466944
Title: Quantitative Magnetic Resonance Imaging of Bone Marrow in a Paediatric Population With Leukaemia (PUMA)
Brief Title: PUMA (Paediatric Osseous Marrow Assessment)
Acronym: PUMA
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor Nandita DeSouza, Principle Investigator (Joint Head of Unit, Radiotherapy & Imaging), Institute of Cancer Research, United Kingdom
Other Study IDs: 18/SW/0021 CCR 4779
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Leukaemia
Keywords: Magnetic Resonance Imaging (MRI); Leukaemia; Whole-Body DiffusionWeighted-Magnetic Resonance Imaging (WB DW-MRI); Paediatrics
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5-24 year old paediatric patients with childhood Leukaemia: Cooperative paediatric individuals and young adults (5-24-years-old) with proven Acute Lymphoblastic Leukaemia (ALL) or Acute Myeloblastic Leukaemia (AML) planned for bone marrow transplantation.

SUMMARY:
This is a pilot cancer imaging study investigating change in the apparent diffusion coefficient (ADC) at a single time point post-transplantation in patients. The treatment is bone marrow transplant as per standard patient care, without change for trial purposes.

Its main aim is to evaluate the engraftment of bone marrow after transplantation performing functional Magnetic Resonance Imaging (MRI) of the lumbar spine and pelvis at baseline and after 2-3 weeks after the transplantation (according to the appearances of raised white blood cells).This will enhance the understanding of bone marrow features on imaging at engraftment and improve the management of children/young adults who suffer acute leukaemia.

Following allogenic haemopoietic stem cell transplantation, changes in bone marrow apparent diffusion coefficient (ADC) are measurable at the point of engraftment and in conjunction with peripheral blood counts may provide a future biomarker of successful clinical outcome.

DETAILED DESCRIPTION:
This is a single-center pilot study. The investigators intend to image 12 inpatients, aged 5-24 years old who are scheduled for haemopoietic stem cell transplantation.

Patients will have two MRI scans requiring them to lie in the scanner for approximately 15 minutes. Patients unable to tolerate lying flat for this length of time or to tolerate the scan for any reason will be withdrawn from the study. If required a play specialist can be organised to help the young patients feel more at ease in the MRI department. MRI does not involve radiation exposure and when performed within national safety guidelines do not pose a significant risk. Patients with contraindications to MRI such as pacemakers, certain metal implants and claustrophobia will not be recruited. Every effort will be made to book scan appointments to coincide with clinic visits.

Scans will be reported as per clinical procedures and data will be made available to the referring consultants immediately via the radiology picture archiving and communications system (PACS).

ELIGIBILITY:
Inclusion Criteria:

1. All patients with relapsed or high risk acute lymphoblastic or myeloblastic leukaemia planned for haemopoietic stem cell transplantation
2. Cooperative paediatric individuals and young adults (5-24-years-old) not requiring general anaesthesia or sedation for the purpose of MRI
3. Able to lie flat throughout the scan

Exclusion Criteria:

1. Non cooperative patients
2. Ferromagnetic implants, contraindicating MRI
3. Claustrophobia
4. Unable to lie flat throughout the scan
5. Uncertain histological diagnosis
6. Musculoskeletal disorders
7. Metabolic disorders
8. Lack of signed parental consent and patient's verbal approval

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A pilot paediatric cohort of 12 patients with Acute lymphoblastic leukaemia (ALL) or Acute myeloid leukemia (AML), aged 5-25 years old, will be studied before and after haemopoietic stem cell transplantation.
  Patients with either of the two types of acute leukaemia will be included.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The change in ADC following bone marrow transplantation at the point of engraftment in paediatric patients with leukaemia. | 8 months
  Measured as the percentage of children who achieve a change in ADC of their bone marrow with engraftment that is greater than the limits of agreement of repeatability of the measurement, established from previous historical data.

SECONDARY OUTCOMES:
Heterogeneity of ADC distribution within lumbar spine & pelvis before and after engraftment, evaluated as the mean ADC. | 8 months
  This will be evaluated for each patient in each scan (mean ADC for each Region Of Interest) and summarised with histograms and descriptive statistics.
Correlation between ADC change and white blood cell count | 8 months
Comparison of baseline ADC between patients with treated ALL and treated AML | 8 months
  A baseline magnetic resonance scan with diffusion-weighted images and without contrast administration will be performed at the end of the neoadjuvant treatment (chemotherapy with/without radiation depending on the type of leukaemia).

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — ICR
Locations (1):
- The Institute of Cancer Research and Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom